CLINICAL TRIAL: NCT03362944
Title: Physiological Correlates of Active Music-making and Passive Listening in Music Based Interventions
Brief Title: Active and Passive Music Therapy Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-2508; 2KR961706 (Other Grant/Funding Number: NCTraCS)
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-03

CONDITIONS: Autonomic Nervous System Imbalance; Hypothalamic Pituitary Adrenal Axis Suppression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Music Therapy (Experimental)
  Interventions: Behavioral: Active Music Therapy
- Passive Music Therapy (Experimental)
  Interventions: Behavioral: Passive Music Therapy

INTERVENTIONS:
Behavioral: Active Music Therapy — The intervention consists of a standardized series of Music Therapy tasks, all based at a constant rhythmic pulse.
  Arms: Active Music Therapy
Behavioral: Passive Music Therapy — The intervention consists of a series of recorded listening tracks, matched in style to the active intervention, all based at a constant rhythmic pulse.
  Arms: Passive Music Therapy

SUMMARY:
Purpose: In this preparatory study, the investigators will demonstrate the feasibility of using a structured MT intervention as a treatment for MDD by measuring stress hormone levels and HRV before and after interventions.

Participants: Participants will be healthy controls ages 18 to 34 years old, both male and female, english speakers, with no history or cardiovascular or neurological diseases.

Procedures: A passive listening control will be used in conjunction with an active music therapy intervention to assess whether the physiological correlates can be targeted by active music-making. Participants will experience both the control and the intervention in separate sessions for a within participants design. HRV and saliva samples will be recorded pre and post intervention for both sessions. The investigators anticipate that the active MT intervention will produce greater physiological changes (pre intervention to post intervention) than the passive listening control. Model-based estimation of treatment effects and components of variance will inform our choice of the sample size deemed necessary for a subsequent grant-funded MT-MDD clinical trial.

DETAILED DESCRIPTION:
Music therapy (MT) interventions are a cost-effective, accessible, and holistic treatment option with social, rhythmic, creative, sensorimotor, and respiratory components, giving them the potential to improve the quality of life for a diverse array of disorders. Despite this, the literature surrounding MT is controversial due to the lack of standardization in clinical and research practice. Interventions range from passive listening of participant selected music to clinician lead improvisational sessions. This inhibits a mechanistic understanding of how MT functions, and what components produce therapeutic effects. Controlled studies that target physiological outcomes are vital for the development of evidence-based MT treatments.

Major depressive disorder (MDD) is a leading cause of disability for U.S. and affects more than 16 million Americans each year. Existing interventions struggle to combat this societal burden and fail to reach the large number of treatment resistant patients, creating an urgent need for the development of new treatment paradigms. Hyperactivity of the hypothalamic-pituitary-adrenal (HPA) axis and dysregulation of the autonomic nervous system (ANS) have been implicated in MDD. Listening to music has been shown to alter stress hormone levels and heart rate variability (HRV), physiological correlates of the HPA axis and ANS respectively. Active music-making's effects on these correlates has yet to be studied. Since active musical engagement involves multiple sensory inputs-proprioceptive and motor in addition to auditory-it has the potential to heighten physiological changes associated with listening to music alone. By contrasting a structured participation MT intervention with a listening control, the investigators will target the effects of active participation in music-making as a potential treatment for MDD.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 34 years of age
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)

Exclusion Criteria:

* Non-English speaker
* Cardiovascular disease
* Neurological diseases
* On medication for cardiovascular or neurological disorders

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill Medical School Wing C, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Rafieyan R, Ries R. A description of the use of music therapy in consultation-liaison psychiatry. Psychiatry (Edgmont). 2007 Jan;4(1):47-52. PMID 20805929
- [Background] Thaut MH, McIntosh GC, Hoemberg V. Neurobiological foundations of neurologic music therapy: rhythmic entrainment and the motor system. Front Psychol. 2015 Feb 18;5:1185. doi: 10.3389/fpsyg.2014.01185. eCollection 2014. PMID 25774137
- [Background] Ellis RJ, Thayer JF. Music and Autonomic Nervous System (Dys)function. Music Percept. 2010 Apr;27(4):317-326. doi: 10.1525/mp.2010.27.4.317. PMID 21197136
- [Background] Linnemann A, Ditzen B, Strahler J, Doerr JM, Nater UM. Music listening as a means of stress reduction in daily life. Psychoneuroendocrinology. 2015 Oct;60:82-90. doi: 10.1016/j.psyneuen.2015.06.008. Epub 2015 Jun 21. PMID 26142566
- [Background] Dean J, Keshavan M. The neurobiology of depression: An integrated view. Asian J Psychiatr. 2017 Jun;27:101-111. doi: 10.1016/j.ajp.2017.01.025. Epub 2017 Jan 29. PMID 28558878
- [Background] Mikutta CA, Schwab S, Niederhauser S, Wuermle O, Strik W, Altorfer A. Music, perceived arousal, and intensity: psychophysiological reactions to Chopin's "Tristesse". Psychophysiology. 2013 Sep;50(9):909-19. doi: 10.1111/psyp.12071. Epub 2013 Jun 14. PMID 23763714
- [Background] Rajendra Acharya U, Paul Joseph K, Kannathal N, Lim CM, Suri JS. Heart rate variability: a review. Med Biol Eng Comput. 2006 Dec;44(12):1031-51. doi: 10.1007/s11517-006-0119-0. Epub 2006 Nov 17. PMID 17111118
- See also: National Institute of Mental Health (2015). Major Depression Among Adults — https://www.nimh.nih.gov/health/statistics/prevalence/major-depression-among-adults.shtml

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were excluded from the study prior to assignment to groups.
Groups:
- Active Music Therapy Followed by Passive Music Therapy: Active Music Therapy: The intervention consists of a standardized series of Music Therapy tasks, all based at a constant rhythmic pulse.
  Passive Music Therapy: The intervention consists of a series of recorded listening tracks, matched in style to the active intervention, all based at a constant rhythmic pulse.
  Interventions were spaced at minimum one week apart.
- Passive Music Therapy Followed by Active Music Therapy: Passive Music Therapy: The intervention consists of a series of recorded listening tracks, matched in style to the active intervention, all based at a constant rhythmic pulse.
  Active Music Therapy: The intervention consists of a standardized series of Music Therapy tasks, all based at a constant rhythmic pulse.
  Interventions were spaced at minimum one week apart.
Period: First Intervention
Arm/Group | Active Music Therapy Followed by Passive Music Therapy | Passive Music Therapy Followed by Active Music Therapy
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Single Week Washout Period
Arm/Group | Active Music Therapy Followed by Passive Music Therapy | Passive Music Therapy Followed by Active Music Therapy
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Active Music Therapy Followed by Passive Music Therapy | Passive Music Therapy Followed by Active Music Therapy
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Includes all participants in both treatment arms:
  * Active Music Therapy followed by Passive Music Therapy
  * Passive Music Therapy followed by Active Music Therapy
  Active Music Therapy: The intervention consists of a standardized series of Music Therapy tasks, all based at a constant rhythmic pulse.
  Passive Music Therapy: The intervention consists of a series of recorded listening tracks, matched in style to the active intervention, all based at a constant rhythmic pulse.
  For each arm interventions were spaced at minimum one week apart.
Arm/Group | Overall Study
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Post Intervention High Frequency (HF) and Low Frequency Divided by High Frequency (LF/HF) Power Amplitude
Description: Five minute heart-rate variability (HRV) recordings will be taken before and after each intervention session through two electrodes placed on the participant's right collarbone and left rib cage. The recordings will be analyzed for HF and LF/HF components, which correspond with sympathetic and parasympathetic autonomic nervous system (ANS) activity.
Time Frame: Before and after 40-minute intervention
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Active Music Therapy | Passive Music Therapy
Number analyzed (Participants) | 16 | 16
Decibels
  HF power | 0.1796 (1.6943) | 0.1507 (0.7360)
  LF/HF power | -0.3872 (0.6961) | 0.3731 (0.7693)

2. Primary Outcome: Change From Baseline to Post Intervention Cortisol
Description: Stress hormone levels correspond with hypothalamic-pituitary-adrenal (HPA) axis activity. This will be assessed using saliva swabs.
Time Frame: Before and after 40-minute intervention
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter
Arm/Group | Active Music Therapy | Passive Music Therapy
Number analyzed (Participants) | 16 | 16
Micrograms per deciliter | -0.0496 (0.0949) | -0.0174 (0.0558)

3. Primary Outcome: Change From Baseline to Post Intervention Alpha-amylase (A-amylase)
Description: Stress hormone levels correspond with HPA axis activity. This will be assessed using saliva swabs.
Time Frame: Before and after 40-minute intervention
Measure: Mean (Standard Deviation); unit: units per milliliter
Arm/Group | Active Music Therapy | Passive Music Therapy
Number analyzed (Participants) | 16 | 16
units per milliliter | -19.0285 (52.2087) | -3.9287 (32.8864)

4. Secondary Outcome: Active and Passive Music Therapy Post Intervention HF and LF/HF Power Amplitude
Description: Post intervention HRV recordings, assessed through two electrodes placed on the participant's right collarbone and left rib cage, will be compared between the Active and Passive intervention conditions.
Time Frame: Interventions are administered 1 week apart, post intervention recordings will be taken and compared on a 1 week time frame.
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Active Music Therapy | Passive Music Therapy
Number analyzed (Participants) | 16 | 16
Decibels
  HF power | 1826 (1723) | 1220 (877.0)
  LF/HF power | 1.344 (1.141) | 1.753 (1.459)

5. Secondary Outcome: Active and Passive Music Therapy Post Intervention Cortisol
Description: Post intervention stress hormone levels, as assessed through saliva swabs, will be compared between the Active and Passive intervention conditions.
Time Frame: Interventions are administered 1 week apart, post intervention stress hormone levels will be assessed and compared on 1 week time frame.
Measure: Mean (Standard Deviation); unit: micrograms per deciliter
Arm/Group | Active Music Therapy | Passive Music Therapy
Number analyzed (Participants) | 16 | 16
micrograms per deciliter | .1784 (.0884) | .1839 (.0902)

6. Secondary Outcome: Active and Passive Music Therapy Post Intervention A-amylase
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units per milliliter
Arm/Group | Active Music Therapy | Passive Music Therapy
Number analyzed (Participants) | 16 | 16
Units per milliliter | 75.02 (62.87) | 57.31 (45.31)

ADVERSE EVENTS:
Time Frame: Collection of adverse events ranged from enrollment to the completion of the second intervention. This time course was approximately 1 month for each participant.
Arm/Group | Active Music Therapy | Passive Music Therapy
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03362944/Prot_SAP_000.pdf